CLINICAL TRIAL: NCT03863379
Title: Sarcopenic Obesity in Neurodisabled People
Brief Title: Sarcopenic Obesity in Neurodisabilities
Acronym: SarcObeNDS
Status: Completed | Type: Observational
Sponsor: Dionyssiotis, Yannis, M.D. (Individual)
Collaborators: University of Athens (Other); University of Patras (Other)
Responsible Party: Principal Investigator, Yannis Dionyssiotis, Consultant of 1st PRM Department National Rehabilitation Center EKA, Athens, Greece, University General Hospital of Patras
Other Study IDs: AFIAP2019-01
Record Dates: First submitted 2019-02-28; First posted 2019-03-05 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Sarcopenic Obesity; Spinal Cord Injuries; Stroke; Multiple Sclerosis; Traumatic Brain Injury
Keywords: Sarcopenia; sarcopenic obesity; stroke; sci; TBI; MS
MeSH Terms: conditions — Spinal Cord Injuries; Stroke; Multiple Sclerosis; Brain Injuries, Traumatic; Sarcopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neurodisabled persons: Persons with various neurodisabilities
  Interventions: Diagnostic Test: whole body DXA
- Control group: Able bodied persons
  Interventions: Diagnostic Test: whole body DXA

INTERVENTIONS:
Diagnostic Test: whole body DXA — Measurements of body composition may be used to study how lean body mass and body fat change during health and disease and have provided a research tool to study the metabolic effects of obesity and various wasting conditions. DXA measurements are based in part on the assumption that the hydration of fat-free mass remains constant at 73%.

SUMMARY:
To describe the frequency and thresholds for sarcopenic obesity in neurodisabled persons and the fat and lean mass distribution based on various neurodisabilities

ELIGIBILITY:
Inclusion Criteria:

Persons with

* stroke / cerebrovascular disease
* traumatic brain injury
* multiple sclerosis
* spinal cord injuries (including spinal cord lesions i.e. myelopathies etc.)

Exclusion Criteria:

Persons with

* heterotopic ossifications,
* chronic administration of drugs, which promote fat increase
* chronic administration of drugs, which promote bone or muscle loss
* co-existing other diseases such as: endocrinopathies, muscular dystrophies, non-alcoholic fatty liver disease.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons with neurodisability, men and women in comparison with able-bodied controls. Controls considered healthy after physical examination and comprehensive medical history review, which was free of any previous fracture ,endocrine or metabolic bone disease, malignancy, drug abuse, alcoholism and hepatic or renal disorders.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Fat and lean mass in neurodisabled | an average of 1 year
Frequency of sarcopenic obesity | an average of 1 year

SECONDARY OUTCOMES:
Body mass index correlation with fat mass and visceral fat | an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- National Rehabilitation Center EKA, Nea Liosia, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kalinkovich A, Livshits G. Sarcopenic obesity or obese sarcopenia: A cross talk between age-associated adipose tissue and skeletal muscle inflammation as a main mechanism of the pathogenesis. Ageing Res Rev. 2017 May;35:200-221. doi: 10.1016/j.arr.2016.09.008. Epub 2016 Oct 1. PMID 27702700
- [Result] Pelletier CA, Miyatani M, Giangregorio L, Craven BC. Sarcopenic Obesity in Adults With Spinal Cord Injury: A Cross-Sectional Study. Arch Phys Med Rehabil. 2016 Nov;97(11):1931-1937. doi: 10.1016/j.apmr.2016.04.026. Epub 2016 Jun 7. PMID 27282328
- [Result] Polyzos SA, Margioris AN. Sarcopenic obesity. Hormones (Athens). 2018 Sep;17(3):321-331. doi: 10.1007/s42000-018-0049-x. Epub 2018 Jul 16. PMID 30014320
- [Derived] Dionyssiotis Y, Prokopidis K, Trovas G, Papadatou MC, Ananidis N, Tragoulias V, Lazarou E, Christaki E, Domazou M, Galanos A, Tyllianakis M. Sarcopenic Obesity in Individuals With Neurodisabilities: The SarcObeNDS Study. Front Endocrinol (Lausanne). 2022 Jul 19;13:868298. doi: 10.3389/fendo.2022.868298. eCollection 2022. PMID 35928890